CLINICAL TRIAL: NCT03679936
Title: Diagnostic Significance of Single Center, Open and Prospective Evaluation of <Sup>18<Sup>F-FDG PET/CT Dynamic Imaging and Genomic Sequencing in Detecting Metastatic Lesions and Differentiating Multiple Primary Lung Cancer From Intrapulmonary Metastases of Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.FZYX.002
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Positron-Emission Tomography; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Biopsy, Needle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — needle biopsy of tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non-metastatic group: PET/CT dynamic scan,needle biopsy and gene detection
  Interventions: Diagnostic Test: PET/CT dynamic scan
- Metastatic group: PET/CT dynamic scan,needle biopsy and gene detection
  Interventions: Diagnostic Test: PET/CT dynamic scan
- Multiple primary lung cancer group: PET/CT dynamic scan,needle biopsy and gene detection
  Interventions: Diagnostic Test: PET/CT dynamic scan
- Intrapulmonary metastases group: PET/CT dynamic scan,needle biopsy and gene detection
  Interventions: Diagnostic Test: PET/CT dynamic scan

INTERVENTIONS:
Diagnostic Test: PET/CT dynamic scan — This study is designed to evaluate the patients who are first diagnosed with non-small cell lung cancer (NSCLC)，for 18 F-FDG PET/CT dynamic scanning and primary tumors and/or metastases in biopsy, than find the inner link of the tumor imaging findings, genomics and histopathologic characteristics, discuss diagnostic value of 18 F-FDG PET/CT dynamic imaging in metastatic non-small cell lung cancer (NSCLC). At the same time, evaluating the ability of 18 F-FDG PET/CT dynamic imaging to differentiating multiple primary lung cancer from intrapulmonary metastases.
  Other Names: Needle biopsy; Gene detection

SUMMARY:
The purpose of this study is to evaluate the diagnostic value of 18F-FDG PET/CT dynamic imaging in metastasis of non-small cell lung cancer (NSCLC). The investigators will collect dynamic 18F-FDG PET/CT scan and correlate the imaging findings with genomics and histopathological features of biopsy of primary or / and metastatic lesions in patients with newly diagnosed non-small cell lung cancer (NSCLC). At the same time, the investigators will evaluate the diagnostic value of 18F-FDG PET/CT dynamic imaging in differentiating multiple primary lung cancer from intrapulmonary metastases.

DETAILED DESCRIPTION:
Lung cancer is a malignant tumor with the highest morbidity and mortality in China and all over the world, in which non-small cell lung cancer (NSCLC) accounts for more than 85% of all categories [1-2]. Although the precision medicine has greatly improved the survival time of patients with NSCLC, most patients still have recurrence and metastasis after a period of time [3]. The nature of tumorigenesis, development and metastasis is a series of biochemical processes, such as abnormal gene expression and metabolism, dysfunction and structural change. Early prediction of tumor metastasis and accurate and timely clinical intervention will not only help clinicians to formulate treatment plans, but also reduce unnecessary side effects and medical expenses with ineffective treatment. 18F-FDG-PET scans can reflect metabolic changes at cellular and molecular level, and the metabolic information are transmitted earlier than anatomical changes. Detection of 18F-FDG uptake, analysis of tumor metabolism, tissue blood flow perfusion, receptor, and so on, can provide a theoretical basis for monitoring the therapeutic efficacy of lung cancer by PET [4].

As a new imaging technique, 18F-FDG PET/CT plays a more and more important role in the diagnosis of tumor. 18F-FDG PET/CT reflects the process of glucose metabolism in tumor tissue. The diagnosis of benign and malignant tumors is based on the difference of glucose metabolism activity between tumor cells and normal tissue cells. 18F-FDG is the isomer of glucose, which participates in the process of glucose metabolism. Because it cannot produce hexose diphosphate because of its deoxidation, it cannot participate in the next metabolism, and it is retained in cells. Due to the high expression of glucose transport mRNA,the level of Glut-1 and Glut-3 increased, the expression of hexokinase increased, and the level of glucose-6-phosphatase decreased, which resulted in an increase of 18F-FDG uptake in tumor cells [5]. Molecular imaging using 18F-FDG PET / CT can provide metabolic information, which can make benign and malignant tissues differentiate better, and reveal the functional abnormalities before structural damage [6]. However, the current PET/CT scans reported in the relevant literature are based on conventional static scans, i.e. the image data is based on a static take-up image of the tracer in tissue obtained at a fixed time point after the injection of 18F-FDG. To improve, the investigators propose to use dynamic data scanning, which captures the dynamic data of whole body tissues collected from the moment of injecting 18F-FDG to an hour. Dynamic scans can provide information on the dynamic changes in tracer metabolism and distribution in tissues over time, so they provide a richer metabolic and distributional pattern of tumor foci and metastases than static scans. Therefore, the aim of this study is to make up for this gap by performing a dynamic scan of 18F-FDG PET/CT on newly diagnosed patients with non-small cell lung cancer. The lesions and/or metastases are performed for biopsy. Pathological and genomic studies are performed. The differences between tumor images and tissues are compared at the same time. 18F-FDG PET/CT dynamic imaging is explored in non-small cell lung cancer metastases for the diagnostic value.At the same time, the ability to differentiate multiple primary lung cancer from intrapulmonary metastases of 18F-FDG PET/CT dynamic imaging will be dissussed .

ELIGIBILITY:
Inclusion Criteria:

* Accurately diagnosing primary liver cancer according to pathological diagnostic criteria or clinical diagnostic criteria.
* Tumor volume (> 1 cm) displayed by enhanced CT or MRI or liver mass confirmed by arteriography .
* For patients considering distant metastases, trunk metastases need to be confirmed by CT examination. Bone metastases need to be confirmed by whole-body bone scan. Brain metastases need to be confirmed with characteristic metastatic tumors by MRI.
* The age is more than 18 years old and less than 65 years old. There is no gender restriction.
* Untreated patients who have not received surgery, interventional therapy, chemotherapy, biotherapy, and radiation therapy.
* Physical condition score ECOG: 0-2; no major organ dysfunction; oxygen partial pressure ≥ 10.64kPa; white blood cell count≥ 4 × 109/L; hemoglobin ≥ 9.5g/dL; neutrophil absolute count ≥ 1.5 × 109 / L; platelet count ≥ 100 × 109 / L; total bilirubin ≤ 1.5 times of the upper limit of normal value; creatinine ≤ 1.25 times of the upper limit of normal value; and creatinine clearance ≥ 60ml / min.
* Be able to obtain complete follow-up information, understand the situation of this study and sign informed consent.

Exclusion Criteria:

* Poorly controlled diabetics (fasting blood glucose levels > 200 mg/dL).
* In addition to four types of malignant tumors that can be treated with radical resection, such as cervical cancer in situ, basal or squamous cell skin cancer, (breast) ductal carcinoma in situ, and organ localized prostate cancer, suffering from any other malignant tumors within 5 years.
* Breastfeeding and/or pregnant women.
* Patients with severe bleeding tendencies (prothrombin time less than 50%, cannot be corrected by treatment with vitamin K, etc.).
* Recent severe hemoptysis, severe cough, dyspnea or patients are not able to cooperate.
* People with severe emphysema, pulmonary congestion, and pulmonary heart disease.
* Researchers believe that the subject may not be able to complete this study or may not be able to comply with the requirements of this study (for management reasons or other reasons).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: More than 18 years old and less than 65 years old, no gender limitation, first diagnosis of non-small cell lung cancer patients, patients who must comply with all the inclusion criteria are eligible to participate in this study.However,patients who meet any of the exclusion criteria will not be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Calculating the overall diagnostic sensitivity and specificity and ROC | 60 minutes
  For each patient enrolled in the study, a two-chamber four-parameter model (2TCM) and a Patlak two-parameter model are established using 18F-FDG PET/CT dynamic scans. Summarizing these dynamic model parameters for all enrolled patients separately calculates the overall diagnostic sensitivity and specificity. Calculate ROC based on sensitivity and specificity.

SECONDARY OUTCOMES:
Calculating the overall diagnostic sensitivity and specificity and summarizing the intrinsic correlation | 60 minutes
  Summarize the genetic testing of all enrolled patients and radiomic indicators to calculate the overall diagnostic sensitivity and specificity. At the same time, the intrinsic correlations between genomics, gene detection and histopathology are summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Hongjun Jin, Zhuhai, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang M, Lin Z, Xu Z, Li D, Lv W, Yang S, Liu Y, Cao Y, Cao Q, Jin H. Influx rate constant of 18F-FDG increases in metastatic lymph nodes of non-small cell lung cancer patients. Eur J Nucl Med Mol Imaging. 2020 May;47(5):1198-1208. doi: 10.1007/s00259-020-04682-5. Epub 2020 Jan 23. PMID 31974680